CLINICAL TRIAL: NCT00429390
Title: Effect of Fasting With Two Meals on Insulin Resistance Indices of Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Free Islamic University of Medical Sciences (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1345103
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2007-01-31 (Estimated); Status verified 2007-01

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic syndrome; Ramadan Fasting; Insulin sensitivity; Iran
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance

INTERVENTIONS:
Behavioral: Ramadan Fasting

SUMMARY:
this study was conducted to assess the insulin resistance indices in the subjects undergoing Ramadan fasting (diet which consisted of two meals at 12 hours intervals)for a thirty days period.

DETAILED DESCRIPTION:
Insulin resistance is a feature of a number of clinical disorders, including type 2 diabetes/glucose intolerance, obesity, dyslipidaemia and hypertension clustering in the so-called metabolic syndrome.The prevalence of the metabolic syndrome, as defined by the 2001 ATP III criteria, was 22 percent, with an age-dependent increase.Data demonstrates that the prevalence has continued to increase, particularly in women.Hyperinsulinemia occurring in response to insulin resistance may play an important role in the genesis of metabolic syndrome. Prevention or reduction of obesity, particularly abdominal obesity, is the main therapeutic goal in patients with the metabolic syndrome .Weight reduction is optimally achieved with a multimodality approach including diet, exercise, and possible pharmacologic therapy, as with orlistat .It has been shown that many different diets such as Mediterranean diet, DASH diet, Foods with low glycemic index and low saturated fat diet, independent of weight loss, by reducing insulin resistance may be effective in improving the metabolic syndrome .During the month of Ramadan (The ninth month of the Islamic calendar), Muslims fast every day from dawn to sunset. They refrain from drinking and eating for about 12h intervals. There are currently no reports on the effect of Ramadan fasting (only two meals per day) on metabolic syndrome. Therefore, this study was conducted to assess the insulin resistance indices in the subjects undergoing this type of fasting for a thirty days period.

ELIGIBILITY:
Inclusion Criteria:

* Males with metabolic syndrome

Exclusion Criteria:

Conditions with insulin resistance including:

* Type 2 diabetes mellitus
* Infections
* Stresses
* Uremia
* Acromegaly
* Glucocorticoid excess
* Hypertension
* Cirrhosis and;
* Any addiction or drug therapy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55
Dates: Start 2006-08; Study Completion 2006-11

PRIMARY OUTCOMES:
Measuring insulin sensitivity in metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Zahra V Shariatpanahi, MD, Principal Investigator — Islamic Free University of Medical Science